CLINICAL TRIAL: NCT04099420
Title: Differences in Behaviour Related to Dietary Habit, Self-medication and Nutraceuticals Use Among Italian and Spanish University Students: Relationship With Cardiovascular Risk Factors.
Brief Title: Lifestyle, Self-medication and Use of Nutraceuticals in a Population of Italian and Spanish Students
Acronym: STANIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maura Palmery (Other)
Collaborators: Universidad Católica San Antonio de Murcia (Other); Research Centre for Food and Nutrition, CREA - AN (Unknown)
Responsible Party: Sponsor-Investigator, Maura Palmery, Associate Professor of Pharmacology, University of Roma La Sapienza
Organization: University of Roma La Sapienza (Other)
Other Study IDs: 1382/2019; CE071906 (Other: Universidad Católica San Antonio de Murcia (UCAM))
Record Dates: First submitted 2019-08-18; First posted 2019-09-23 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Medication Adherence
Keywords: Self-medication; Adherence to Mediterranean diet; Orthorexia; Relationship lifestyle and metabolic status biomarkers; Oral microbiota composition; Relationship lifestyle and immunological status biomarkers
MeSH Terms: conditions — Medication Adherence; Orthorexia Nervosa

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — The urine will be collected by the volunteers through the common sterile containers and data normalized for creatinine, after control with urine strip (11 parameters).
  After delivery, the saliva and urinary samples will be frozen and transported to the Center of Food Research and Nutrition (CREA-AN) for subsequent analysis.
  The composition of the oral microbiota will be evaluated through genomic DNA extraction from a salivary sample and subsequent Next Generation Sequencing analysis of the 16S ribosomal deoxyribonucleic acid (rDNA).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Italian university students: university students, doctoral students, post-docs and post-graduate students in biomedical and pharmaceutical sciences (N = 100)
  Interventions: Behavioral: Lifestyle counseling
- Spanish university students: university students, doctoral students, post-docs and post-graduate students in biomedical and pharmaceutical sciences (N = 100)
  Interventions: Behavioral: Lifestyle counseling

INTERVENTIONS:
Behavioral: Lifestyle counseling — An in-depth analysis of the lifestyle of Italian and Spanish university students will be carried out for the first time, with assessment of the frequency of self-medication and use of drugs and supplements/nutraceuticals. The composition of the oral microbiota in relation to eating habits will be determined for the first time. The results of this study will be useful for designing promotion programs for the correct use of drugs/supplements and for healthy diets and lifestyles in university students

SUMMARY:
University students are considered a population class with a high risk of malnutrition and/or obesity, metabolic and cardiovascular diseases, with a tendency to misuse drugs and self-medication.

The interest in a healthy diet can lead to a psychological obsession known as orthorexia, frequent among students in the biomedical field and in the sports context.

The high levels of stress recorded in university students have been related to the use of drugs to enhance their cognitive abilities. The phenomenon of self-medication is one of the main problems for public health, with high levels recorded among students of health professions.

A high adherence to the Mediterranean diet seems to bring health benefits, with an impact even on the intestinal microbiota composition. Although several studies have investigated the effect of the Mediterranean diet on intestinal microbiota, little attention has been paid to the effect of this diet on the oral microbiota, one of the most relevant microbial habitats from a clinical point of view.

The aim of this study is to evaluate self-medication, adherence to the Mediterranean diet, the relationship between lifestyle and biomarkers of the metabolic and immunological status, and impact of eating habits on the oral microbiota composition.

Students, doctoral students, post-docs and specialists in the biomedical and pharmaceutical fields will be recruited in Italy (N = 200) and in Spain (N = 200). Data will be collected through questionnaires in order to evaluate self-medication, eating habits, level of physical activity, orthorexia and lifestyle of the subjects. The entire group will be evaluated with clinical parameters of metabolic status and the quality of saliva and urine. The latter will be determining factors for the selection of 50 Italian and 50 Spanish students, on which parameters of immunological and antioxidant status, cortisol, urinary phenols, and the composition of the oral microbiota will be evaluated.

Italian and Spanish students may have different eating habits and lifestyles. It is assumed that subjects with high adherence to the Mediterranean diet have a better metabolic and immunological status. Moreover, high rates of orthorexia are expected among students who practice sports. The composition of the oral microbiota could vary depending on the type of diet and consistently with the immunological status markers.

DETAILED DESCRIPTION:
Young people are considered a population at risk of nutritional deficiencies due to bad eating habits, found especially among university students. In fact, the latter tend to change their eating habits when they begin their university studies, with adherence to a typically western diet that includes low consumption of fish, fruit and vegetables, monounsaturated and polyunsaturated fatty acids, and an increase in consumption of sugars, alcohol and "fast food", with the consequent increase in this population class of the risk of malnutrition and/or obesity, metabolic and cardiovascular diseases. These changes are due to the lack of experience in meal planning, with a consequent increase in the frequency of meals away from home, to the increase in the number of snacks or meals skipped to respect the timetable of the lessons, to the easier access to the fast food and limited economic resources. Among the unhealthy behaviors adopted by the students, in addition to the wrong eating habits, there are also reduced physical activity, increased sedentariness, alcohol consumption and smoking.

Over the past 20 years there has been an increase in obesity rates among university students who, especially for medical students, are closely related to specific habits such as: skipping breakfast, attending fast food, low fruit and vegetables consumption, and easy access to unhealthy foods from the machines. Among the freshmen, especially those who live far from families and find themselves independent for the first time in their lives, higher rates of weight gain and higher levels of stress have been reported, responsible for changes in food choices. In fact, to control stress levels, individuals are encouraged to prefer foods that are high in fat. Therefore, university students should be seen as a group that requires special attention regarding health promotion, especially food.

However, the interest in a healthy diet can lead to a psychological obsession known as orthorexia (ortho = just, oreksis = appetite), which consists in the persistent concern of maintaining the self-imposed diet to improve one's health. Nutritionists/dieticians and students are the categories of population most affected by orthorexia, with a prevalence in Italian nutrition science students of 35.9%. The typical behaviors of orthorexia can be associated with a negative image of one's own body, despite the subject's strong interest in appropriate and healthy food choices. However, as a result of extreme restriction/concern over one's diet, orthorhexics would tend to eliminate whole groups of foods with consequent nutritional deficiencies, malnutrition and weight loss. Furthermore, the typical eating behavior of orthoressia is associated with intense physical activity, suggesting that students who practice sports have a greater tendency to develop this disorder.

The high levels of stress recorded in university students were also related to the use of smart drugs and "smart nutrients", which university students, especially those in medicine (74.7%), use to enhance their cognitive abilities. The phenomenon of self-medication is one of the main problems for public health, with only 48% of the population of the European Union using prescribed drugs. Among the students of health professions high levels of self-medication with antibiotics are recorded in the absence of indication. Another trend that is of particular concern is the increase in the use of antidepressants among young people, which many of them take after disappointments in academic performance and which have negative side effects such as weight gain , altered lipid profile and risk of diabetes. Another category of substances that young people abuse or otherwise misuse are amphetamines, and the co-intake of stimulants, alcohol or other drugs is also of concern. Indeed, a recent study carried out on Italian and Spanish pharmacy students showed that Spaniards have a high percentage of drug use and that 38.4% of subjects take them in conjunction with alcohol; instead, Italian students have revealed that they rarely turn to the pharmacist and rely more on the advice of family or friends.

The university years therefore represent a period marked not only by food problems but also by stress, anxiety, depression and other psychological problems. However, it emerged that a high adherence to the Mediterranean diet would bring benefits at the cognitive level, with an improvement in the states of depression and anxiety and a better academic result. In addition to a healthy diet, even moderate and regular physical activity (90 minutes a week) has been shown to reduce levels of anxiety and depression with improved well-being and self-esteem. For this reason it is essential to promote this lifestyle among university students.

Different types of diet and bioactive compounds taken with the diet can also have an impact on the composition of the intestinal microbiota. In particular, the Mediterranean diet has been associated with a greater abundance of Bacteroidetes, Prevotellacea and Prevotella and a lower concentration of Firmicutes and Lachnospiraceae. Although several studies have investigated the eating habits of Spanish university students, only Scuri et al. investigated the use of drugs in Italian and Spanish university students, but limited the study to a well-defined sample represented by students of the only pharmacy faculty, because they were considered particularly careful and involved on this topic. It would therefore be interesting to evaluate this behaviour, including the tendency to self-medication, between Italian and Spanish students, including biomedical and not just pharmaceutical faculties, in order to have an overview of the behaviour of university students who support scientific studies, that should lead them to acquire more awareness of health problems, including the correct use of drugs. Furthermore, although several studies have investigated the effect of the Mediterranean diet on intestinal microbiota, little attention has been paid to the effect of this diet on the oral microbiota, despite the oral cavity being one of the most relevant microbial habitats from a clinical point of view, and it has been shown to be a significant risk factor for cardiovascular diseases, diabetes mellitus, bacteraemia and tumors. It is therefore interesting to analyse and investigate these aspects.

The aim of this study is to evaluate self-medication, adherence to the Mediterranean diet, the relationship between lifestyle and biomarkers of the metabolic and immunological status, and impact of eating habits on the oral microbiota composition.

Primary goals:

* Compare the prescription of drugs and the use of alcohol, energy drinks, supplements, dietary products and/or other types of nutraceuticals in Italian and Spanish university students.
* Compare the adherence to the Mediterranean diet in Italian and Spanish university students.
* Compare cardiovascular risk factors (obesity, hypertension, hyperglycemia, dyslipidemia and smoking habits) and ketosis in Italian and Spanish university students.

Secondary goals:

* Compare and evaluate the level of physical activity and the percentage of subjects with orthorexia nervosa in Italian and Spanish university students.
* Compare the frequency and type of meals consumed outside home, the type and consumption of food/beverages and adherence to special dietary regimes (vegetarian diet, ketogenic etc), in Italian and Spanish university students.
* Register other characteristics of interest (pathologies, anxiety/depressive symptoms, food neophobia, eating disorders, vaccinations and opinion on vaccines).
* Compare eating habits, salivary microbiota and salivary immunoglobulin A (IgA), interleukin-6 (IL-6) and cortisol levels in a sub-group of non-smoking Italian and Spanish students.

In the recruitment phase it will be sent to the subjects by e-mail:

* "The" INFORMATION NOTE AND CONSENT "
* "Food Diary" (optional completion)

From the time of recruitment to enrolling (first meeting) the volunteers will be able to calmly and carefully read the "INFORMATION AND CONSENT NOTE". The subjects may also request clarifications or details from the recruiter and/or the person in charge of the study. Moreover, before deciding, the volunteers will have time to ask an opinion to family or to a doctor of their trust.

The recruiters will make contact with the volunteers, collect the data and assign a code to the volunteer.

The standard data flow at the first, second and third meeting will be as follows:

First meeting:

1. Signed informed consent at the time of enrollment.
2. Compilation of the "Code sheet"
3. Withdrawal and control of the "food diary"
4. Filling in questionnaires
5. Anthropometric and arterial pressure measurements

Second meeting:

1. New notice of the information note and informed consent signature
2. Administration of the Food Frequency Questionnaire (FFQ) (http://www.sisdca.it/public/pdf/IDAO---testistica.pdf) with the aid of the Scotti Bassani portant atlas (http: // www .giorgiobedogni.it / archives / text / atlas / patlante.html)
3. Collection of saliva samples to assess their quality and for subsequent analysis
4. Delivery container for collection of urine and those for the collection of saliva for circadian cortisol.

Third meeting:

1. New notice of the information note and informed consent signature
2. Delivery of urine and saliva samples collected
3. Measurement of metabolic state parameters (cholesterol, triglycerides, glycemia and ketones)

An in-depth analysis of the lifestyle of Italian and Spanish university students will be carried out for the first time, with assessment of the frequency of self-medication and use of drugs and supplements/nutraceuticals. The composition of the oral microbiota in relation to eating habits will be determined for the first time. This study should also confirm the results of previous studies on the high rate of orthorexia in biomedical faculty students, especially among nutritionists and sports practitioners. The results of this study will also be useful for designing promotion programs for the correct use of drugs/supplements and for healthy diets and lifestyles in university students, and will also provide a potentially useful basis for the recruitment of subjects in additional/future intervention studies.

ELIGIBILITY:
Inclusion Criteria:

* university students, doctoral students, post-docs and post-graduate students in biomedical and pharmaceutical sciences

Exclusion Criteria:

* age <18 years or inability to sign informed consent.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: University students, doctoral students, post-docs and post-graduate students in biomedical and pharmaceutical sciences (N = 200, 100 Italian and 100 Spanish).
  The sample size was chosen based on previous studies conducted on university students. If no significant differences were found for the markers for which there is no supporting literature, the sample size will be calculated for subsequent studies, setting a desidered power 0.8 with an alpha = 0.05, based on the average difference and the standard deviation of the compared groups (Italian and Spanish students in relation to the degree of adherence to the Mediterranean diet)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-07-17 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Compare the prescription of drugs in Italian and Spanish university students | One year
  The percentage of subjects who resort to self-medication and the use of drugs will be evaluated on the basis of the data reported in a specific online questionnaire
Compare the use of alcohol in Italian and Spanish university students | One year
  The use of alcoholic beverages will be evaluated with the questionnaire AUDIT, which will be included in the questionnaire on "voluptuous habits"
Compare the use of energy drinks in Italian and Spanish university students | One year
  The use of energy drinks will be evaluated on the basis of the data reported in a specific online questionnaire
Compare the use of supplements, dietary products and/or other types of nutraceuticals in Italian and Spanish university students | One year
  The use of supplements, dietary products and / or other types of nutraceuticals will be evaluated on the basis of the data reported in a specific online questionnaire
Compare the adherence to the Mediterranean diet in Italian and Spanish university students | One year
  The degree of adherence to the Mediterranean diet (online questionnaire) will be calculated with two different scores: the Mediterranean Diet Score (MDS) evaluated through the validated 14-item questionnaire of the PREDIMED study and the MEDScore (Score-55) proposed by Panagiotakos with the dedicated software. The latter, unlike the first, includes the consumption of unrefined cereals. We will compare the baseline characteristics of participants according to three categories of adherence to the Mediterranean diet (> or egual to 5, 6-9 and > or egual to 10 points of the 14-item questionnaire). At each question of the 14-item questionnaire will be assigned a score of 0 or 1 on the basis of the answer. Panagiotakos et al. have already proposed a diet score that evaluates adherence to the Mediterranean diet through a large-scale (from 0 to 55).
Compare cardiovascular risk factors (obesity) in Italian and Spanish university students | Two year
  Measurements of weight (Kg), height (m) (portable mechanical Stadiometer), lean mass and fat mass will be recorded on the data collection form. In particular, the latter will be measured both by means of the OMRON BF-511 body analysis impedance balance and by plicometry. Weight and height will be combined to report BMI in kg/m^2
Compare cardiovascular risk factors (hypertension) in Italian and Spanish university students | Two year
  Blood pressure will be recorded on the data collection form
Compare cardiovascular risk factors (hyperglycemia and dyslipidemia) in Italian and Spanish university students | Two year
  The clinical metabolic status parameters will be evaluated by: self-diagnosis of capillary blood sampling (cholesterol, triglycerides and glycaemia by means of Multicare IN) and a dedicated ELISA kit for saliva sample insulin, based on saliva quality.
Compare ketosis in Italian and Spanish university students | Two year
  The clinical metabolic status parameter will be evaluated by self-diagnosis of capillary blood sampling (ketones by means of ON Call GK Dual)

SECONDARY OUTCOMES:
Compare and evaluate the level of physical activity in Italian and Spanish university students | One year
  The level of physical activity will be evaluated using the International Physical Activity Questionnaire (IPAQ, online questionnaire). It covers four domains of physical activity: work-related, transportation, housework/gardening and leisure-time activity. The questionnaire also includes questions about time spent sitting as an indicator of sedentary behaviour. In each of the four domains the number of days per week and time per day spent in both moderate and vigorous activity are recorded. At work, during transportation and in leisure time, walking time is also included. Moderate intensity is defined as 3-6 MET (Metabolic Equivalent Task) and vigorous intensity was defined as >6 MET. One MET is equal to energy expenditure during rest and is approximately equal to 3.5 ml O2 kg^-1 min^-1 in adults.
Compare and evaluate the percentage of subjects with orthorexia nervosa in Italian and Spanish university students | One year
  The frequence of orthorexia nervosa will be evaluated using the ORTO-15 test (online questionnaire).Answers that indicate orthorexia are given a score of "1", while the "healthier" ones have a score of "4". The sum of the scores is the final score of the test. We set a threshold value of 40. Below this cut-off the test is supposed to give a diagnosis of orthorexia.
Compare the frequency of meals consumed outside home in Italian and Spanish university students | One year
  Outcome Measure will be evaluated by online questionnaires
Compare the type of meals consumed outside home in Italian and Spanish university students | One year
  Outcome Measure will be evaluated by online questionnaires
Compare the type of food/beverages consumed in Italian and Spanish university students | One year
  Outcome Measure will be evaluated by online questionnaires
Compare the consumption of food/beverages in Italian and Spanish university students | One year
  Outcome Measure will be evaluated by online questionnaires
Compare the adherence to special dietary regimes (vegetarian diet, ketogenic etc) in Italian and Spanish university students | One year
  Outcome Measure will be evaluated by online questionnaires
Register other characteristics of interest (pathologies) | One year
  Other characeristics of interest will be evaluated by online questionnaires
Register other characteristics of interest (anxiety/depressive symptoms) | One year
  Other characeristics of interest will be evaluated by online questionnaires
Register other characteristics of interest (food neophobia) | One year
  Other characeristics of interest will be evaluated by online questionnaires
Register other characteristics of interest (eating disorders) | One year
  Other characeristics of interest will be evaluated by online questionnaires
Register other characteristics of interest (vaccinations and opinion on vaccines) | One year
  Other characeristics of interest will be evaluated by online questionnaires
Compare eating habits in a sub-group of non-smoking Italian and Spanish students | Two year
  Eating habits will be evaluated by online questionnaires
Compare salivary microbiota in a sub-group of non-smoking Italian and Spanish students | Two year
  The composition of the oral microbiota will be evaluated through genomic DNA extraction from a salivary sample and subsequent Next Generation Sequencing analysis of the 16S rDNA.
Compare salivary IgA levels in a sub-group of non-smoking Italian and Spanish students | Two year
  Salivary IgA levels will be measured with ELISA kit
Compare salivary IL-6 levels in a sub-group of non-smoking Italian and Spanish students | Two year
  Salivary IL-6 levels will be measured with ELISA kit
Compare salivary cortisol levels in a sub-group of non-smoking Italian and Spanish students | Two year
  Salivary cortisol levels will be measured with ELISA kit

CONTACTS AND LOCATIONS:
Overall Officials: Maura Palmery, Professor, Study Director — La Sapienza University of Rome, Italy
Locations (3):
- Italy (2):
  - Research Centre for Food and Nutrition, Council for Agricultural Research and Economics (CREA-AN), Rome
  - La Sapienza University, Rome
- Universidad Catolica San Antonio de Murcia, Murcia, Guadalupe, Spain

IPD SHARING:
Plan to Share IPD: Yes
The study will be articulated both in Italy and in Spain as follows:
  2019-2020 phase Italy 2020-2021 phase Spain 2022 end of the study 2019-2022 publications and congresses